CLINICAL TRIAL: NCT06396832
Title: POST-SURGICAL SYMPTOMS IN PATIENTS UNDERGOING GASTRIC SLEEVE SURGERY: OMENTOPEXY VS. NO OMENTOPEXY
Brief Title: Comparing Post-Surgical Symptoms: Gastric Sleeve With and Without Omentopexy "Comparing Post-Surgical Symptoms: Gastric Sleeve With and Without Omentopexy" Comparison of Postoperative Symptoms: Gastric Sleeve With and Without Omentopexy.
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: OMENTOPEXY-2024
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Omentopexy; Complications; Metabolic surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing gastric sleeve surgery with omentopexy: Omentopexy aims to prevent or reverse sleeve gastrectomy complications, but it is not a standardized technique by itself, with more than 5 descriptions of it. Among the authors who have presented their technique are Sharma, Batman, Pilone, Abou Ashour, Nosrati, and Labib. It consists of fixing the remnant stomach with the gastrosplenic and gastrophrenic ligaments to stabilize the posterior aspect of the stomach and prevent gastric torsion, a functional cause of stenosis
- Patients undergoing conventional sleeve gastrectomy: The procedure is associated with other complications, some of which are believed to be related to loss of fixation of the stomach to the greater omentum. Among the main ones is nausea, exacerbation or onset of symptoms due to reflux, as well as intolerance to certain foods and regurgitation

SUMMARY:
Metabolic surgery has proven to be an effective treatment for obesity, with laparoscopic sleeve gastrectomy being the most popular procedure. Omentopexy (OP) is proposed as a strategy to reduce associated complications. Objective was to determine the effectiveness of omentopexy in controlling post-surgical symptoms and to measure the need for re-intervention, leakage, bleeding, and mortality in patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Patients who underwent laparoscopic sleeve gastrectomy (LSG). Of these patients, 53 received LSG with omentopexy (OP) and 52 underwent LSG without omentopexy (NO OP) between 2022 and 2023. Each group was attended by a different surgeon. The analysis focused on data concerning gastrointestinal symptoms recorded 24 hours postoperatively, as well as documented cases of bleeding, leakage, re-operation, and mortality during the hospitalization period

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity
* Adults over 18 years old
* Undergoing sleeve gastrectomy
* Consent to respond to the immediate postoperative symptom questionnaire

Exclusion Criteria:

* Repair of hiatal hernia
* Refusal to complete the evaluation instrument
* Unavailability of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with obesity who underwent sleeve gastrectomy, with or without omentopexy
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative gastrointestinal symptoms | 24 hours
  patients undergoing sleeve gastrectomy with omentopexy for obesity treatment will be lower compared to those undergoing sleeve gastrectomy without adjuncts.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, Mexico, Guadalajara, Jalisco, Mexico